CLINICAL TRIAL: NCT01485731
Title: Phase 1 Study of Nelfinavir Added to Cisplatin Chemotherapy Concurrent With Pelvic Radiation for Locally Advanced Cervical Cancer (II-IVA)
Brief Title: Safety Study of Nelfinavir + Cisplatin + Pelvic Radiation Therapy to Treat Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Matt Pearson, Assistant Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20100153
Record Dates: First submitted 2011-11-29; First posted 2011-12-05 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Cervical Cancer
Keywords: Cervical; Cancer; Uterine Cervix; Squamous Cell; Adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms; Adenocarcinoma | interventions — Nelfinavir; Cisplatin; Brachytherapy; Papanicolaou Test; Hearing; Proctoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nelfinavir + Cisplatin + Pelvic Radiation Therapy (Experimental): Nelfinavir in combination with Cisplatin and Pelvic Radiation Therapy
  Interventions: Drug: Nelfinavir; Drug: Cisplatin; Radiation: Pelvic External Beam Radiation Therapy; Radiation: Brachytherapy; Procedure: Pharmacokinetic Sampling; Procedure: Cervical Biopsy; Procedure: Pelvic Examination; Procedure: Pap Smear; Procedure: Audiogram; Procedure: Proctoscopy; Procedure: Cytoscopy; Procedure: Renal Ultrasound; Procedure: CT Scan; Procedure: Whole Body PET/CT Scan

INTERVENTIONS:
Drug: Nelfinavir — Nelfinavir (NFV) will be prescribed orally twice daily for 7 days prior to initiation of cisplatin and pelvic radiation at the starting dose level, 875 mg BID
  Other Names: NFV
Drug: Cisplatin — Cisplatin at 40 mg/m2 (maximum total dose of 70 mg per week), will be infused intravenously once per week on either Day 1, 2, 3, 4, or 5 of weeks 2 to 6, preferably approximately four hours prior to radiation therapy. One additional cycle of cisplatin will be given either week 7 or 8 for a total of 6 cycles of cisplatin. Patients are not to be dosed more than 70 mg/week.
Radiation: Pelvic External Beam Radiation Therapy — Pelvic external beam radiation therapy (PEBRT) will be delivered in combination with weekly IV cisplatin (40mg/mg2) and twice daily oral NFV.PEBRT should be delivered once each day during the business week (Monday to Friday) according to the acceptable standards of care as prescribed by the treating radiation oncologist(s). The radiation therapy should consist of whole pelvic external beam radiation therapy (WPEBRT) with or without a parametrial boost (PB). PEBRT will be interdigitated with one administration of intrauterine brachytherapy (BT) given on any business day of week 7 or 8.
  Other Names: PEBRT
Radiation: Brachytherapy — PEBRT will be interdigitated with one administration of intrauterine brachytherapy (BT) given on any business day of week 7 or 8.
  Other Names: BT
Procedure: Pharmacokinetic Sampling — Serum levels of Nelfinavir will be assayed at the following 3 time points: 5-8 days after initiation of NFV single agent (on Day 5, 6, or 7 of week 1 or day 1 of week 2), 1 week after combined NFV and cisplatin pelvic radiation (on day 15, 16, or 17 if start on Monday) for measurement of steady state, and at the completion of treatment (within the last 3 days of radiation in week 6). Blood samples will be taken before drug administration on the day of the sample to make sure the concentrations are actually at a minimum and before tumor biopsies.
Procedure: Cervical Biopsy — Three punch biopsies of cervical tumor will be obtained during office visit at each time point (for PCR, IHC, and banked for future research). NFV serum levels will be obtained once NFV has been started (day 5-8 pre chemoradiation and at completion of chemoradiation) before each cervical biopsy
Procedure: Pelvic Examination — Pre-Treatment, at the end of treatment +/- 1 week, every 3 months +/- 2 weeks after therapy (x 1 year)
Procedure: Pap Smear — Recommended. Every 3 months +/- 2 weeks after therapy (x 1 year)
Procedure: Audiogram — Required in patients with history of hearing loss; 28 days within starting treatment and every other cycle.
Procedure: Proctoscopy — Optional. Pre-Treatment
Procedure: Cytoscopy — Optional. Pre-Treatment
Procedure: Renal Ultrasound — Optional. Pre-Treatment
Procedure: CT Scan — CT Scan of Chest/Abdomen/Pelvis, pre-treatment,Immediately at end of trial +/- 1 week, Every 3 months +/- 2 weeks after therapy (x 1 year)
Procedure: Whole Body PET/CT Scan — In lieu of CT Scan, pre-treatment,Immediately at end of trial +/- 1 week, Every 3 months +/- 2 weeks after therapy (x 1 year)

SUMMARY:
Nelfinavir will increase the efficacy of Cisplatin based chemo- radiation therapy for locally advanced cervical cancer.

DETAILED DESCRIPTION:
Despite cisplatin chemoradiation, 40-50% of women with locally advanced cervical cancer will die from their disease. The evaluation of new chemoradiation regimens have since included cisplatin to further build on its current success. In one year, Nelfinavir will be off patent and become a potential cost effective therapy. HIV Protease inhibitors are now being explored as potential therapies in oncology. The repositioning of HIV protease inhibitors, specifically nelfinavir in cancer therapeutics, is based on three facts. First, recent studies show that HIV protease inhibitors are established broad-spectrum anti-cancer agents that work through pleiotropic mechanisms such as by down-regulating activated mitogenic signaling pathways, and activating the immune response with Nelfinavir being the most potent [7]. Second, HIV protease inhibitors including nelfinavir can target specific viral antigens. Nelfinavir has been shown to target Human Papilloma Virus (HPV)-transformed cervical carcinoma cells via inhibition of E6-mediated proteosomal degradation of mutant p53 [8]. Thirdly, Nelfinavir has radiosensitizing properties through inhibiting the PI3K/Akt signaling pathway as demonstrated in vivo and in vitro in head and neck and pancreatic cancers models [9].

Nelfinavir is currently being evaluated as a radiosensitizer in head and neck and pancreatic cancers in phase I/II clinical trials. Brunner et al. (2008) recently completed the first phase I trial of nelfinavir added to chemoradiation for locally advanced pancreatic cancer [16]. Investigators treated 12 patients with advanced pancreatic carcinoma with Nelfinavir 1250 mg orally twice daily starting 3 days before radiation therapy and continued until the last day of radiation. They found no significant toxicity attributable to nelfinavir and observed a response rate of 50% versus 30% in historical controls. There were 5 of 12 patients with grade 3 hematologic toxicities (4 with leukopenia and 2 with thrombocytopenia). There were 3 of 12 patients with grade 3 GI toxicity (including abdominal pain, nausea, vomiting). There were no grade 4 drug related toxicities [16]. There were grade 1/ 2 toxicities including hematologic (thrombocytopenia, anemia, neutropenia), gastrointestinal toxicities (nausea, vomiting, diarrhea, abdominal pain), and elevated transaminases which were approximately 70%. Ten of 12 patients completed therapy. Complete responses were observed in 5 patients and partial responses were observed in 5 of 10 patients. Overall, the addition of Nelfinavir added minimal additional toxicity. Determination of a dose for biologic activity was not performed [14].

In summary, HIV protease inhibitors have a very broad spectrum of anti-tumor activity and can inhibit proliferation and/or cause death in the majority of cancer cell lines tested in a dose-dependent manner [7]. Nelfinavir has been found to be the most potent anti-tumor agent among the HIV protease inhibitors. As a result, several clinical trials are investigating Nelfinavir as a chemotherapeutic agent with and without concurrent radiation therapy in varied disease sites including rectal, head & neck, glioblastomas, pancreas, renal cell, non-small cell lung cancer, liposarcoma, and gliomas. The NCI is also investigating Nelfinavir as single agent chemotherapy in advanced and recurrent solid tumors [15].

As Nelfinavir has both cytotoxic and radiation sensitizing effects, it is an ideal agent to use in combination with cisplatin-based chemoradiation in locally advanced cervical cancers.

In this study, patients with clinical stages IIA, IIB, IIIA, IIIB, IVA cervical carcinoma limited to the pelvis will receive twice daily oral Nelfinavir (NFV) and weekly IV cisplatin in combination as radiosensitizers with daily whole pelvic external beam (Mon-Fri) followed by intracavitary radiation brachytherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary, previously untreated, histologically confirmed invasive carcinoma of the uterine cervix (any cell type). Clinical stages IIA, IIB, IIIA, IIIB, IVA.
* Patients must have adequate bone marrow, renal and hepatic function:

  * ANC ≥ 1,500/μL;
  * Platelet count ≥ 100,000/μL;
  * Creatinine < 2.0 mg/dL;
  * Total Bilirubin ≤ 1.5 times normal;
  * SGOT ≤ 3 times normal.
* Patients with a GOG Performance Status of 0, 1, or 2.
* Patients with ureteral obstruction must be treated with stent or nephrostomy tube.
* Patients must be entered within eight weeks of diagnosis.
* Patients of childbearing potential must use an effective form of birth control."Patients receiving oral contraceptives should be instructed that alternate or additional contraceptive measures should be used during therapy with VIRACEPT. "
* Seronegative HIV status.
* Patients must be at least 18 years of age.
* Patients must have signed an approved informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

* Patients with Stage IA, IB or IVB disease.
* Patients who have known metastases to other organs outside the radiation field at the time of the original clinical and surgical staging.
* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy.
* Patients with septicemia or severe infection.
* Patients who have circumstances that will not permit completion of this study or the required follow-up.
* Patients who are pregnant at the time of diagnosis and do not wish pregnancy termination prior to initiation of treatment.
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields.
* Patients with other concomitant malignancies (with the exception of non-melanoma skin cancer), who had (or have) any evidence of other cancer present within the last 5 years.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Patients with poorly controlled diabetes mellitus despite medication.
* Patients taking anti-arrhythmic agents such as amiodarone, quinidine, rifampin, ergot derivatives such as ergotamine, St Johs Wort, HMG-CoA reductase inhibitors such as lovastatin, neuroleptic such as pimozide, sedatives such as midazolam and triazolam among other CYP3A4 and CYP2C19 substrates.
* Patients with Phenylketonuria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Adverse Events in Phase 1 Study of Nelfinavir + Cisplatin + Pelvic Radiation Therapy | 3 Years
  Number of Patients with Adverse Events in Phase 1 Study of Nelfinavir + Cisplatin + Pelvic Radiation Therapy
The proportion of enrolled patients for whom Nelfinavir dose can be successfully administered in combination with Cisplatin and Pelvic Radiation Therapy. | 3 Years
  Maximum tolerable Phase II dose of Nelfinavir in combination with Cisplatin and Pelvic Radiation Therapy.

SECONDARY OUTCOMES:
Serum Levels of Nelfinavir and other Biomarker Activity | 3 Years
  To determine the levels of Akt activity (and downstream effectors such as pGSK3, pEBP1) and p16INK4A in addition to the presence of Human Papilloma Virus (HPV) 16 and18,and E6/E7 RNA in cervical biopsy specimens of patients at three different time points (1. pre-nelfinavir, pre-radiation, 2. while on nelfinavir, pre-radiation, 3. at completion of radiation therapy), and correlate the levels of these markers to serum Nelfinavir levels from blood drawn at the day of the biopsy.
Response to protocol therapy | 3 years
  Tumor response to protocol therapy will be measured using Response Evaluation Criteria In Solid Tumors (RECIST) criteria.
Progression-free Survival | 3 years
  Progression-Free Survival is the period from start of treatment until documented disease progression or death from any cause. For surviving patients without progression, progression-free survival will be censored at the last date of documented progression-free status.
Overall Survival | 3 years
  Survival is the observed length of life from start of treatment to death. For surviving patients, follow-up will be censored at the date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: J. Matthew Pearson, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States